CLINICAL TRIAL: NCT05574283
Title: Erector Spinae Plane Block Versus Quadratus Lumborum Block for Postoperative Analgesia After Laparoscopic Resection of Colorectal Cancer: A Prospective Randomized Study
Brief Title: Erector Spinae Plane Block Versus Quadratus Lumborum Block for Postoperative Analgesia After Laparoscopic Resection of Colorectal Cancer.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Hebatullah Negm Eldeen Abd El Azeem, lecturer of anaesthesia, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMBSUREC/11092022/Negm
Record Dates: First submitted 2022-10-04; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESPB group (Experimental): ESPB group: 30 patients will receive bilateral ultrasound-guided erector spinae plane block using 20 ml of bupivacaine 0.25% with 4 mg dexamethasone for each side.
  Interventions: Procedure: Erector spinae plane block and transmuscular quadratus lumborum block
- TQLB group (Experimental): TQLB group: 30 patient will receive bilateral ultrasound-guided transmuscular quadratus lumborum block using 20 ml of bupivacaine 0.25% with 4 mg dexamethasone for each side.
  Interventions: Procedure: Erector spinae plane block and transmuscular quadratus lumborum block

INTERVENTIONS:
Procedure: Erector spinae plane block and transmuscular quadratus lumborum block — All blocks were performed after securing the airway before the start of surgery.
  ESPB group will receive bilateral ultrasound-guided erector spinae plane block using 20 ml of bupivacaine 0.25% with 4 mg dexamethasone for each side.
  TQLB group will receive bilateral ultrasound-guided transmuscular quadratus lumborum block using 20 ml of bupivacaine 0.25% with 4 mg dexamethasone for each side

SUMMARY:
Colorectal cancers are one of the leading causes of cancer-related mortality, and the incidence is increasing day by day. For this reason, colorectal cancer surgery and postoperative analgesia have gained more importance in recent years.Although laparoscopic surgery is less invasive, it can still generate moderate to severe acute postoperative pain.For a long time, opioids have played a major role in postoperative analgesia, but heavy use of these drugs will cause adverse reactions such as nausea, vomiting and enteroparalysis, which is not conducive to rapid recovery after surgery Therefore, it is critical to developing a more effective regional analgesic technique for patients undergoing abdominal surgery . Erector spinae plane block (ESPB) is a novel interfascial plane block technique that was firstly described in 2016. It involves injecting local anesthetic into the plane between the deep fascia of the erector spinae muscle and the vertebral transverse process under ultrasound guidance to relieve pain in the thoracoabdominal region .The quadratus lumborum block (QLB) is a new posterior abdominal trunk block which produces analgesic effects through local anesthetic that covers thoracolumbar fascia and thoracic paravertebral space. Based on the injection position and approach, there are 3 QLB techniques: lateral approach, posterior approach and anterior approach. The anterior transmuscular quadratus lumborum block (TQLB) is a truncal block (ventral rami of T7- L2) that produces its analgesic effect by blocking the thoracic sympathetic trunk, the ventral rami of lower spinal nerves, the sympathetic fibers and mechanoreceptors within the thoracolumbar fascia, and the celiac ganglion by spread via the splanchnic nerves .

DETAILED DESCRIPTION:
The study will be carried out at Beni-Suef university hospital, after approval by the department of Anesthesiology, Surgical Intensive Care and Pain management, faculty of medicine, Beni-Suef University. The study will be done from october 2022 for 1 year.

Setting: Beni-Suef University Hospital Participants: Eligible patients are aged 35-75 years, with an American Society of Anesthesiologists (ASA) physical status of I-III, and are scheduled to undergo laparoscopic resection of colorectal cancer. Patients willing to participate in the study will get information bedside, and written informed consent will be obtained. Recruitment can of course always be retracted before, during, or even after trial start and will have no influence on further treatment of patient. here is no anticipated harm and compensation for trial participation.

Intervention: All blocks were performed after securing the airway before the start of surgery.

ESPB group will receive bilateral ultrasound-guided erector spinae plane block using 20 ml of bupivacaine 0.25% with 4 mg dexamethasone for each side.

TQLB group will receive bilateral ultrasound-guided transmuscular quadratus lumborum block using 20 ml of bupivacaine 0.25% with 4 mg dexamethasone for each side.

Anesthetic technique:

All the patients will be underwent routine preoperative check-ups, routine haematological and biochemical analyses, and cardiac evaluation. The study protocol will be explained to all participants, including the visual analogue scale (VAS), which will be explained on the day of the preoperative evaluation. Standard monitoring will be established when patients were transferred to the operating room. Invasive arterial blood pressure monitoring, central venous catheter placement right jugular internal vein, and catheterization in the right neck will be performed. patient will receive midazolam 0.05 mg/kg IV 3 minutes prior to induction and ondansetron 4 mg IV. Anaesthesia will be induced by 2-2.5 mg/kg propofol, 2 μg/kg fentanyl & 0.5 mg/kg atracurium for muscle relaxation. The patient will be ventilated using a face mask with 100% oxygen at a rate of 4 L/min and isoflurane 1.2 %. After 180 s, the patient will be intubated using an appropriately sized cuffed oral tube. Anaesthesia maintenance will be performed by isoflurane 1.2% in 100 % O2 and intravenous fentanyl infusion at a rate of 1-2 μg/kg/hr. Muscle relaxation will be continued by atracurium 0.1 mg/kg every 20 min. Mechanical ventilation will be performed for all participants to maintain end-tidal carbon dioxide levels between 35-40 mmHg. Intravenous fluid requirements will be assessed and provided to patients perioperatively, and normothermia will be maintained throughout the procedure. At the end of surgery, a reversal of the muscle relaxant will be done using neostigmine (0.04 mg/kg) and atropine (0.015 mg/kg). After extubation, all patients will be transmitted to the post anesthesia care unit (PACU). When patients were found to be fully awake and vitally stable, they will be transferred to surgical intensive care unit.

The following will be recorded:

* Patients' characteristics: Age, sex, BMI, ASA physical status.
* Time needed to perform technique (min): which was defined as the time needed for adequate ultrasonic visualization, needle introduction, and drug injection (time from placement of ultrasound probe on the patient's skin to the end of local anesthetic injection) .
* Duration of anesthesia, duration of surgery & duration of PACU stay.
* Heart rate (HR), mean arterial blood pressure (MAP), were measured at baseline before induction of anesthesia and then continuously monitored and recorded every 10 min intraoperatively, but recorded at baseline, immediately after induction, at 20 min, 40 min, 1h, 2h after induction and finally at the end of surgery.
* Number of blocked dermatomes: were assessed after recovery of anesthesia using pinprick and cold loss sensation with iced solutions.
* Visual analogue scale (VAS) : was assessed at rest and during movement at 30 min, 1, 3, 6, 12, 24 h postoperatively. A score ≤ 3 was considered acceptable for pain relief. Supplementary rescue analgesia was administered in the form of nalbuphine IV 0.15 mg/kg (at VAS ≥ 4).
* 1st time to rescue analgesic (min): is the time to ask for the first postoperative analgesia (nalbuphine), and was calculated from the end of operation to patient reporting VAS ≥ 3.
* Total dose of rescue analgesia (nalbuphine) (primary outcome), that was consumed in the first 24 h postoperatively.
* Quality of Recovery (QoR)-15 questionnaire scores preoperatively and 24 h postoperatively [using the Korean version of the Quality of Recovery-15 scale ], which can be divided into two components: physical and mental well-being
* Intraoperative and postoperative complications related to the blocks as local anesthetic toxicity, needle injury to essential organs, retroperitoneal hematoma, hypotension, lower limb weakness, . . . etc
* The incidence and severity of postoperative complications, such as hypotension, bradycardia, respiratory depression, sedation, nausea, and vomiting, during the first 24 h postoperative were also recorded. A categorical scoring system (0 = none, 1 = nausea, 2 = retching, and 3 = vomiting) was used to evaluate nausea and vomitin . Sedation scores were evaluated using a sedation scale (0 = awake, 1 = drowsy, 2 = asleep but arousable, 3 = deeply asleep). Patients were considered sedated if they had a sedation score of > 0 at any time during the first 24 hours after surgery . Patient satisfaction was assessed as (1 = poor, 2 = moderate, 3 = good, and 4 = perfect) .

ELIGIBILITY:
Inclusion Criteria:

* age between 35 and 75 years.
* patient scheduled for laparoscopic resection of colorectal cancer.
* American Society of Anesthesiologists classification of physical status < IV.
* body's mass index (BMI) ≤ 35 kg/m2.

Exclusion Criteria:

* Refusal of the patient.
* known hypersensitivity to any study medication.
* Chronic opioid use or chronic pain patient.
* Liver insufficiency (defined as a serum bilirubin ≥ 34 μmol/l, albumin ≤ 35 g/dl, INR ≥ 1.7).
* Renal insufficiency (defined as a glomerular filtration rate < 44 ml/min).
* MOrbid obesity (defined as a BMI > 35 kg/m2).
* Obstructive sleep apnea syndrom.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-04 (Actual); Primary Completion 2023-10-04 (Estimated); Study Completion 2023-10-04 (Estimated)

PRIMARY OUTCOMES:
Total dose of rescue analgesia that was consumed in the first 24 hours postoperatively. | First 24 hours postoperatively. Starting immediately after surgery up to 24 hours.
  Total dose of rescue analgesia (nalbuphine) , that was consumed in the first 24 hours postoperatively,if patient visual analogue score more than or equal 3.

SECONDARY OUTCOMES:
1st time to rescue analgesic (min). | First 24 hours postoperatively. Starting from the end of the surgery up to 24 hours..
  It is the time to ask for the first postoperative analgesia (nalbuphine), and was calculated from the end of operation to patient reporting VAS ≥ 3.

CONTACTS AND LOCATIONS:
Overall Officials: hebatullah Negmeldeen, lecturer, Principal Investigator — Beni-Suef University
Locations (1):
- Benisuef university, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Mahmoud Fakhry D, ElMoutaz Mahmoud H, Yehia Kassim D, NegmEldeen AbdElAzeem H. Erector Spinae Plane Block versus Quadratus Lumborum Block for Postoperative Analgesia after Laparoscopic Resection of Colorectal Cancer: A Prospective Randomized Study. Anesthesiol Res Pract. 2024 Mar 18;2024:6200915. doi: 10.1155/2024/6200915. eCollection 2024. PMID 38529324